CLINICAL TRIAL: NCT01826279
Title: Short-term Investigation of Resveratrol on Lipid Turnover in Morbidly Obese Women Undergoing Gastric Bypass Surgery. Effects on Basal and Insulin Stimulated FFA and VLDL-triglyceride Metabolism and Liver VLDL-triglyceride Uptake.
Brief Title: Short-term Investigation of Resveratrol on Fat Metabolism in Morbidly Obese Women Undergoing Gastric Bypass Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: M-20110172B
Record Dates: First submitted 2013-04-03; First posted 2013-04-08 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2013-05

CONDITIONS: Obesity
Keywords: Obesity; Gastric bypass surgery; Resveratrol; Insulin sensitivity; Lipid turnover; VLDL-triglyceride uptake; Liver
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resveratrol (Experimental): Resveratrol 500mg 3 times daily for 1 month
  Interventions: Dietary Supplement: Resveratrol
- Placebo (Placebo Comparator): Placebo 1 tablet 3 times daily for 1 month
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol — 500mg 3 times daily for 1 month
  Arms: Resveratrol
Other: Placebo — 1 placebo tablet 3 times daily for 1 month
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate potential metabolic effects of resveratrol in morbidly obese women undergoing gastric bypass surgery.

The investigators hypothesize that resveratrol will:

* Decrease hepatic very-low-density-lipoprotein-triglyceride (VLDL-TG) secretion
* Decrease hepatic and adipose tissue VLDL-TG uptake
* Increase insulin sensitivity

The investigators will look at changes in:

* Lipid turnover (VLDL-TG kinetics, palmitate kinetics,calorimetry)
* VLDL-TG uptake in different tissues (subcutaneous femoral adipose tissue, subcutaneous abdominal adipose tissue, visceral adipose tissue and liver tissue)
* Insulin sensitivity (glucose kinetics during hyperinsulinaemic euglycaemic clamp)
* Regulation of liver fat handling
* Lipoprotein lipase activity and fat cell size (abdominal and femoral adipose tissue)

ELIGIBILITY:
Inclusion Criteria:

* Female
* 25-60 years
* Obesity (BMI > 35 kg/m2)
* Have at least one element of the metabolic syndrome either hypertension and/or hypercholesterolemia (high triglyceride, low HDL-cholesterol)
* Undergoing gastric bypass surgery
* Written informed consent

Exclusion Criteria:

* Any other relevant disease (e.g. diabetes, thyroid or parathyroid disease, heart, kidney or liver disease)
* May have arthrosis or depression
* Any present or previous malignancy
* History of smoking
* Alcohol dependency (more than 14 units of alcohol per week)
* Participation in studies with radioactive isotope within the last six months
* Hemoglobin under the normal range regarding to sex (under 7.3 mmol/l for women)

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Hepatic VLDL-TG secretion and peripheral VLDL-TG clearance | 1 month
  - changes from baseline after treatment with either resveratrol or placebo
Hepatic and adipose VLDL-TG uptake | 1 month
  - changes in VLDL-TG uptake in resveratrol group and placebo group

SECONDARY OUTCOMES:
Basal and insulin stimulated free fatty acid (FFA) and glucose turnover | 1 month
  - changes from baseline after treatment with either resveratrol or placebo
VLDL-TG oxidation | 1 month
  - changes from baseline after treatment with either resveratrol or placebo
Regulation of liver fat handling | 1 month
  - changes in regulation of liver fat handling in resveratrol group and placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Søren Nielsen, MD, associate professor, DMSc, Study Chair — Department of Endocrinology and Internal Medicine
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus C, Denmark